CLINICAL TRIAL: NCT03235102
Title: Obesity ACTION Study in Canada
Brief Title: Awareness, Care and Treatment in Obesity Management
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-4411; U1111-1199-1902 (Other: World Health Organization (WHO))
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- People with Obesity: People with obesity, or weight loss patients. Potential respondents will be recruited from various Internet patient panels to participate in a cross-sectional, online survey.
  Interventions: Other: No treatment given
- Healthcare Providers: PCPs will include family practitioners; general practitioners; internal medicine; nurse practitioners; and dietitians. Specialists will include endocrinologists and bariatric surgeons, and any of the above if they focus on obesity treatment. Potential respondents will be recruited from various Internet patient panels to participate in a cross-sectional, online survey.
  Interventions: Other: No treatment given
- Employers: Employers in Canada. Potential respondents will be recruited from various Internet patient panels to participate in a cross-sectional, online survey.
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Completion of a survey

SUMMARY:
This study aims to assess barriers that prevent obesity patients from receiving adequate care for their condition. The non-interventional study will be administered in the form of a 30-minute, cross-sectional, online survey to various respondents. There is no experimentation involved in the process of data collection, and each survey poses minimal human risk.

The study will evaluate lifestyle habits and weight management strategies perceived and/or practiced by each of 3 stakeholders in obesity: Patients (People with obesity), Providers, and Employers. A customized survey will be administered to each of the 3 stakeholders, and data will be analyzed based on respondents' answers.

ELIGIBILITY:
Inclusion criteria

The following inclusion criteria will be imposed for HCPs:

* Practice in Canada
* Spends at least 70% of time in direct patient care
* Seen at least 100 patients in past month
* Seen at least 10 patients in past month needing weight management
* In practice 2-35 years
* Not affiliated with Pharmaceutical, Market Research (MR) or Advertising Firms
* PCP - Physician, RN / NP / LPN, or PA, Dietitians
* PCP - Specialty is FP, IM, GP
* Obesity Specialist - Physician, RN / NP / LPN, or PA
* Obesity Specialist - Specialty is FP, IM, GP, endocrinology, bariatrics, or bariatric surgery
* Obesity Specialist - Currently practice as an obesity medicine or weight loss management specialist

The following inclusion criteria will be imposed for PwOs (people with obesity):

* Age at least 18 years
* Lives in Canada
* Recruitment will target a nationally representative Canada sample. Demographic indicators will be monitored throughout recruitment.
* Current BMI 30 kg/sqm or greater, not extremely fit/body building
* Sub-category - Maintaining weight loss: Lost at least 10% of body weight in the past 3 years and has kept weight off for at least a year
* Sub-category - Treatment Seeking: Has committed to a plan to lose weight, or has successfully lost weight (self-report) or has spoken to an HCP about weight loss plan in the last 6 months.

The following inclusion criteria will be imposed for employers:

* Age at least 18 years
* Works in a Canadian province
* Company offers health insurance
* Responsible for making or influencing decisions about health insurance or health and wellness programs
* Works in a company that has 20 or more employees
* Believes there is a weight issue (attitudinal agreement)
* Not affiliated with Pharmaceutical, Market Research (MR) or Advertising Firms

Exclusion criteria Any respondent who work works for a pharmaceutical, health insurance, research, or advertising company will be excluded; as there may be self-presentation effects that could alter the interview questions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All respondents will be recruited from the OMR Globus healthcare panel (http://www.omrglobus.com/). The OMR Globus panel is an opt-in panel, in which respondents join with the understanding they would complete periodic surveys. Members of this panel are not associated with any specific site or organization. Recruitment of these respondents is based on voluntary participation; invitations are sent to the personal e-mail accounts of each respondent.
Sampling Method: Non-Probability Sample
Enrollment: 2545 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
Awareness associated with the care and management of obesity among people with obesity, clinicians and employers | From the first interview on day 1 until the last interview on day 30
  Cross-sectional 30-minute online survey of lifestyle habits and weight management conducted among stakeholders in obesity (clinicians, employers and people with obesity)

CONTACTS AND LOCATIONS:
Locations (1):
- Novo Nordisk Investigational Site, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Sharma AM, Belanger A, Carson V, Krah J, Langlois MF, Lawlor D, Lepage S, Liu A, Macklin DA, MacKay N, Pakseresht A, Pedersen SD, Ramos Salas X, Vallis M. Perceptions of barriers to effective obesity management in Canada: Results from the ACTION study. Clin Obes. 2019 Oct;9(5):e12329. doi: 10.1111/cob.12329. Epub 2019 Jul 11. PMID 31294535